CLINICAL TRIAL: NCT02338882
Title: Randomised Clinical Investigation of the Bi Flex M Multifocal Intraocular Lens
Brief Title: Clinical Investigation of the Bi Flex M Multifocal IOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Phillip J Buckhurst (Other)
Collaborators: BMI Southend Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr Phillip J Buckhurst, Associate Professor (Senior Lecturer), University of Plymouth
Organization: University of Plymouth (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC001
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Cataract
Keywords: Lenses; Intraocular
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bi flex M multifocal intraocular lens (Experimental): Subjects implanted bilaterally with the Bi flex M multifocal intraocular lens
  Interventions: Device: Bi flex M multifocal intraocular lens
- Bi flex 1.8 monofocal intraocular (Active Comparator): Subjects implanted bilaterally with the Bi flex 1.8 monofocal intraocular lens
  Interventions: Device: Bi flex 1.8 monofocal intraocular lens

INTERVENTIONS:
Device: Bi flex M multifocal intraocular lens — Multifocal intraocular lens
  Arms: Bi flex M multifocal intraocular lens
Device: Bi flex 1.8 monofocal intraocular lens — Standard monofocal intraocular lens
  Arms: Bi flex 1.8 monofocal intraocular

SUMMARY:
During cataract surgery an artificial lens is implanted in the eye. These artificial lenses are called intraocular lenses (IOLs) and there are many different types of IOL designs. IOLs are of fixed focus and so unless a multifocal IOL is used you would need to wear spectacles for viewing near objects. This study has been designed to look at how well a multifocal IOL corrects distance and near vision in comparison with a conventional monofocal IOL. Both types of IOLs are commercially available and are commonly implanted. Using new non-invasive methods we hope to be able to better judge the visual performance of these IOLs. In addition the study will involve imaging and examining the IOLs to determine the prevalence of any post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Age related cataract patients requiring cataract surgery with phacoemulsification.
* Patients requiring primary IOL implantation
* Patients with a potential corrected visual acuity of 20/40 or better on clinical assessment
* Patients with normal anterior segments apart from cataracts
* Subjects with clear intraocular media other than cataract

Exclusion Criteria:

* Preexisting pathology or physiology, which may be aggravated by the implant, or may render the implant ineffective and that could potentially cause future acuity losses to a level of 0.5 or 20/40 or worse in either eye. This includes the following:
* Microphthalmia
* Corneal decompensation or Endothelial Insufficiency
* Pseudo exfoliation
* High myopia
* Pars planitis
* Patient with greater than 1 dioptre of preoperative corneal astigmatism
* Subjects who are expected to require retinal laser treatment
* Previous intraocular and/or corneal surgery
* History of uveitis, glaucoma, proliferative diabetic retinopathy, pseudoexfoliation, macular degeneration that may affect potential best corrected visual acuity of 20/40 or better
* Operative complications of posterior capsular rupture, zonular dehiscence, incomplete continuous curvilinear capsulorhexis, severe iris /corneal trauma and inability to achieve secure placement in the designated location
* Subjects using a systemic medication that is known to cause ocular side effects
* Subjects participating in a concurrent clinical trial or if they have participated in an ophthalmology clinical trial within the last 30 days
* Subjects who have only one eye with potentially good vision
* Patients who are not willing to cooperate for the follow up period
* Visual eccentricity of greater than 0.7mm
* Pregnant women
* Patients where it is not possible to take informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip J Buckhurst, PhD, Principal Investigator — Plymouth University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bi Flex M Multifocal Intraocular Lens | Bi Flex 1.8 Monofocal Intraocular
Started | 50 | 50
Completed | 43 | 47
Not Completed | 7 | 3
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Bi Flex M Monofocal Intraocular Lens: Subjects implanted bilaterally with the Bi flex 1.8 monofocal intraocular lens
  Bi flex 1.8 monofocal intraocular lens: Standard monofocal intraocular lens
- Total: Total of all reporting groups
Arm/Group | Bi Flex M Monofocal Intraocular Lens | Bi Flex M Multifocal Intraocular Lens | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (6.4) | 76.6 (6.1) | 76.6 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 39 | 71
  Male | 18 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 50 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50 | 50 | 100
Pupil Size [Mean (Standard Deviation); unit: Millimeters] | 3.72 (0.53) | 3.75 (0.62) | 3.73 (0.57)
Mean Spherical Equivalent [Mean (Standard Deviation); unit: Dioptres] — Manifest refraction performed at distance. Values are for the mean spherical equivalent (MSE) measured in dioptres MSE=sph+(cyl/2)
  Note no changes are necessary
  Dioptres | 0.09 (2.02) | -0.44 (2.42) | -0.17 (2.21)
J0 [Mean (Standard Deviation); unit: Dioptres] — Cylindrical correction defined in vector format. J0 describes astigmatic power along the horizontal meridian
  Dioptres | 0.61 (0.77) | 0.65 (0.69) | 0.62 (.73)
J45 [Mean (Standard Deviation); unit: Dioptres] — Cylindrical correction defined in vector format. J45 describes astigmatic power along the vertical meridian
  Dioptres | 0.02 (0.45) | 0.04 (0.50) | 0.03 (0.47)
Pre-operative corrected distance visual acuity [Mean (Standard Deviation); unit: LogMAR] — Pre-operative best distance corrected visual acuity measured in LogMAR
  LogMAR
    Oculus Dexter (OD) | 0.32 (0.12) | 0.36 (0.14) | 0.34 (0.13)
    Oculus Sinister (OS) | 0.32 (0.13) | 0.36 (0.16) | 0.34 (0.15)

OUTCOME MEASURES:

1. Primary Outcome: Long Term Monocular Visual Acuity (VA)
Description: Monocular Visual acuity at 12-18 months assessed at distance intermediate and near both corrected and uncorrected. Assessed in LogMAR
Time Frame: Visit 2 [12-18 months]
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
LogMAR
  Monocular Uncorrected Distance VA | 0.192 (0.156) | 0.205 (0.138)
  Monocular Uncorrected Near VA | 0.614 (0.198) | 0.319 (0.107)
  Monocular Corrected Distance VA | 0.070 (0.105) | 0.093 (0.090)
  Monocular Distance Corrected Intermediate VA | 0.421 (0.180) | 0.389 (0.130)
  Monocular Distance Corrected Near VA | 0.605 (0.133) | 0.288 (0.143)

2. Primary Outcome: Long Term Binocular Visual Acuity (VA)
Description: Binocular Visual acuity at 12-18 months assessed at distance intermediate and near both corrected and uncorrected. Assessed in LogMAR
Time Frame: Visit 2 [12-18 months]
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Bi Flex M Multifocal Intraocular Lens | Bi Flex 1.8 Monofocal Intraocular
Number analyzed (Participants) | 43 | 47
LogMAR
  Binocular Uncorrected Distance VA | 0.102 (0.100) | 0.093 (0.092)
  Binocular Uncorrected Near VA | 0.275 (0.103) | 0.574 (0.178)
  Binocular Corrected Distance VA | 0.039 (0.070) | 0.031 (0.785)
  Binocular Distance Corrected Intermediate VA | 0.354 (0.103) | 0.393 (0.165)
  Binocular Distance Corrected Near VA | 0.241 (0.100) | 0.571 (0.137)

3. Primary Outcome: Monocular Visual Acuity (VA)
Description: Monocular Visual acuity at 3-6 months assessed at distance intermediate and near both corrected and uncorrected. Assessed in LogMAR
Time Frame: Visit 1 [3-6 months]
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
LogMAR
  Monocular Uncorrected Distance VA | 0.171 (0.144) | 0.183 (0.156)
  Monocular Uncorrected Near VA | 0.576 (0.211) | 0.276 (0.160)
  Monocular Corrected Distance VA | 0.052 (0.083) | 0.076 (0.077)
  Monocular Distance Corrected Intermediate VA | 0.417 (0.134) | 0.393 (0.125)
  Monocular Distance Corrected Near VA | 0.571 (0.180) | 0.271 (0.132)

4. Primary Outcome: Binocular Visual Acuity (VA)
Description: Binocular Visual acuity at 3-6 months assessed at distance intermediate and near both corrected and uncorrected. Assessed in LogMAR
Time Frame: Visit 1 [3-6 months]
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
LogMAR
  Binocular Uncorrected Distance VA | 0.085 (0.105) | 0.101 (0.085)
  Binocular Uncorrected Near VA | 0.554 (0.197) | 0.231 (0.125)
  Binocular Corrected Distance VA | 0.012 (0.072) | 0.044 (0.064)
  Binocular Distance Corrected Intermediate VA | 0.391 (0.128) | 0.378 (0.132)
  Binocular Distance Corrected Near VA | 0.535 (0.170) | 0.236 (0.131)

5. Primary Outcome: Defocus Curve Profiles
Description: Visual acuity measurement (assessed in LogMAR) taken with differing levels of optical defocus
Time Frame: visit 1 (3-6 months)
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
LogMAR
  +1.50 | 0.376 (0.145) | 0.429 (0.139)
  +1.00 | 0.218 (0.093) | 0.300 (0.285)
  +0.50 | 0.089 (0.071) | 0.124 (0.078)
  0.00 | 0.017 (0.072) | 0.050 (0.078)
  -0.50 | 0.104 (0.090) | 0.135 (0.078)
  -1.00 | 0.253 (0.147) | 0.287 (0.101)
  -1.50 | 0.369 (0.167) | 0.328 (0.116)
  -2.00 | 0.505 (0.174) | 0.256 (0.132)
  -2.50 | 0.611 (0.181) | 0.201 (0.180)
  -3.00 | 0.700 (0.169) | 0.235 (0.164)
  -3.50 | 0.745 (0.153) | 0.366 (0.187)
  -4.00 | 0.805 (0.122) | 0.515 (0.149)
  -4.50 | 0.848 (0.113) | 0.610 (0.124)
  -5.00 | 0.893 (0.123) | 0.743 (0.122)

6. Primary Outcome: Long Term Defocus Curve Profiles
Description: Assessed as a dioptric range and using the Defocus area metric
Time Frame: visit 2 (12-18 months)
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
LogMAR
  1.50 | 0.377 (0.150) | 0.359 (0.100)
  1.00 | 0.225 (0.126) | 0.223 (0.089)
  0.50 | 0.093 (0.084) | 0.108 (0.067)
  0.00 | 0.029 (0.082) | 0.043 (0.073)
  -0.50 | 0.111 (0.010) | 0.128 (0.077)
  -1.00 | 0.244 (0.121) | 0.259 (0.085)
  -1.50 | 0.349 (0.159) | 0.309 (0.151)
  -2.00 | 0.499 (0.170) | 0.196 (0.141)
  -2.50 | 0.596 (0.186) | 0.155 (0.113)
  -3.00 | 0.647 (0.171) | 0.188 (0.107)
  -3.50 | 0.692 (0.166) | 0.312 (0.111)
  -4.00 | 0.748 (0.146) | 0.454 (0.118)
  -4.50 | 0.778 (0.127) | 0.563 (0.116)
  -5.00 | 0.804 (0.100) | 0.673 (0.095)

7. Secondary Outcome: Long Term Monocular Pelli-Robson Contrast Sensitivity (CS)
Description: MonocularContrast sensitivity assessed as a contrast threshold using the Pelli-Robson test
Time Frame: Visit 2 [12-18 months]
Measure: Mean (Standard Deviation); unit: Log CS
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
Log CS | 1.347 (0.154) | 1.259 (0.150)

8. Secondary Outcome: Long Term Binocular Pelli-Robson Contrast Sensitivity (CS)
Description: Binocular Contrast sensitivity assessed as a contrast threshold using the Pelli-Robson test
Time Frame: Visit 2 [12-18 month]
Measure: Mean (Standard Deviation); unit: Log CS
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
Log CS | 1.434 (0.136) | 1.379 (0.131)

9. Secondary Outcome: Pelli-Robson Monocular Contrast Sensitivity
Description: Monocular Contrast sensitivity assessed as a contrast threshold using the Pelli-Robson test
Time Frame: Visit 1 [3-6 months]
Measure: Mean (Standard Deviation); unit: Log CS
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 48 | 46
Log CS | 1.428 (0.124) | 1.309 (0.156)

10. Secondary Outcome: Pelli-Robson Binocular Contrast Sensitivity
Description: Contrast sensitivity assessed as a contrast threshold using the Pelli-Robson test
Time Frame: Visit 1 [3-6 months]
Measure: Mean (Standard Deviation); unit: Log CS
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 48 | 46
Log CS | 1.506 (0.088) | 1.391 (0.131)

11. Secondary Outcome: Long Term Contrast Sensitivity CSV-1000
Description: Binocular Assessment of Contrast Sensitivity at threshold using the Contrast sensitivity vision(CSV) CSV-1000
Time Frame: Visit 2 [12-18 months]
Measure: Mean (Standard Deviation); unit: Log CS
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
Log CS
  3 cycles per degree (cpd) | 1.558 (0.162) | 1.515 (0.172)
  6cpd | 1.704 (0.200) | 1.636 (0.161)
  12cpd | 1.379 (0.219) | 1.258 (0.249)
  18cpd | 0.911 (0.216) | 0.765 (0.230)

12. Secondary Outcome: Contrast Sensitivity CSV-1000
Description: Binocular Assessment of Contrast Sensitivity at threshold using the CSV-1000
Time Frame: Visit 1 [3-6 months]
Measure: Mean (Standard Deviation); unit: Log CS
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 48 | 46
Log CS
  3cpd | 1.569 (0.175) | 1.471 (0.180)
  6cpd | 1.771 (0.213) | 1.624 (0.152)
  12cpd | 1.417 (0.261) | 1.249 (0.260)
  18cpd | 0.942 (0.162) | 0.828 (0.261)

13. Secondary Outcome: Long Term Reading Performance
Description: Assessed as the critical print size and using the reading performance index. Uses Radner reading chart and logarithmic Radner scale (LogRAD) Lower LogRAD equals smaller print size
Time Frame: Visit 2 (12-18 months)
Measure: Mean (Standard Deviation); unit: LogRAD
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
LogRAD | 0.948 (0.428) | 0.604 (0.307)

14. Secondary Outcome: Reading Performance
Description: Assessed as the critical print size and using the reading performance index Logarithmic Radner scale (LogRAD) Lower LogRAD equals small print size
Time Frame: visit 1 (3-6 months)
Measure: Mean (Standard Deviation); unit: LogRAD
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
LogRAD | 0.837 (0.297) | 0.692 (0.534)

15. Secondary Outcome: Long Term Glare
Description: Assessed as the glare area size Scale 0 to 100 Higher scores = larger glare area =worse outcome
Time Frame: Visit 2 (12-18 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bi Flex M Monofocal Intraocular Lens | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
units on a scale | 3.78 (14.2) | 37.4 (26.6)

16. Secondary Outcome: Glare
Description: Assessed as the glare area size Scale 0 to 100 Higher score = larger area = worse outcome
Time Frame: visit 1 (3-6 months)
Population: Scale 0 to 100 Higher score = larger glare area = worse outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bi Flex M Monofocal Intraocular Lens | Bi Flex M Multifocal Intraocular Lens
Number analyzed (Participants) | 47 | 43
units on a scale | 4.4 (16.5) | 41.7 (29.4)

ADVERSE EVENTS:
Time Frame: Data collected for 18 months post surgery
Arm/Group | Bi Flex 1.8 Monofocal Intraocular | Bi Flex M Multifocal Intraocular Lens
All-Cause Mortality (participants affected / at risk) | 0/50 | 1/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT02338882/Prot_SAP_000.pdf